CLINICAL TRIAL: NCT01012037
Title: 12 Week Randomised Double-blind BI 1356 2.5 mg Bid vs 5 mg qd add-on to Metformin
Brief Title: Linagliptin 2.5 mg Twice Daily Versus 5 mg Once Daily as add-on Therapy to Twice Daily Metformin in Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.62; 2009-013549-27 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Results first posted 2011-10-31 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

ARMS (3):
- linagliptin low dose (Experimental): linagliptin low dose twice daily
  Interventions: Drug: linagliptin low dose
- placebo (Placebo Comparator): placebo matching linagliptin
  Interventions: Drug: placebo
- linagliptin medium dose (Experimental): linagliptin medium dose once daily
  Interventions: Drug: linagliptin medium dose

INTERVENTIONS:
Drug: linagliptin low dose — patient to receive tablets containing low dose linagliptin twice daily
  Arms: linagliptin low dose
Drug: placebo — patient to receive placebo tablet(s) matching linagliptin
  Arms: placebo
Drug: linagliptin medium dose — patient to receive a tablet containing medium dose linagliptin once daily
  Arms: linagliptin medium dose

SUMMARY:
The objective of the study is to investigate the efficacy and safety of linagliptin 2.5 mg twice daily compared to 5 mg once daily compared to placebo given orally for 12 weeks as add-on therapy to metformin in patients with type 2 diabetes mellitus with insufficient glycaemic control. It is planned to show non-inferiority of linagliptin 2.5 mg twice daily compared to 5 mg once daily and each treatment's superiority over placebo.

ELIGIBILITY:
Inclusion criteria

1. Diagnosis of type 2 diabetes mellitus.
2. Current treatment with metformin alone (>/= 1500 mg or maximally tolerated dose) or metformin plus 1 other antidiabetic drug. Metformin must be administered in twice daily dosing regimen. Patients taking metformin three times daily can be included if posology is switched to twice daily and total daily dose is maintained.
3. Glycosylated haemoglobin (HbA1c) is between 7.0% - 10.0%.
4. Body Mass Index (BMI) </=45 kg/m2.

Exclusion criteria

1. Treatment with extended release metformin.
2. Uncontrolled hyperglycaemia (fasting plasma glucose > 240 mg/dL or 13.3 mmol/L).
3. Myocardial infarction (MI), stroke or transient ischaemic attack (TIA) within 6 months prior to informed consent.
4. Impaired hepatic or renal function, or gastric bypass surgery.
5. Treatment with glitazones, glucagon like peptide-1 (GLP-1) analogues/mimetics, antiobesity agents, or insulin within 3 months of informed consent.
6. Current treatment with systemic steroids or change in dosage of thyroid hormones.
7. Alcohol or drug abuse within 3 months of informed consent.
8. Participation in another trial with investigational drug within 2 months prior to informed consent.
9. Pre-menopausal women who are nursing, pregnant or not practicing an acceptable method of birth control.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (84):
- Belgium (8):
  - 1218.62.32003 Boehringer Ingelheim Investigational Site, De Pinte
  - 1218.62.32008 Boehringer Ingelheim Investigational Site, Kortenaken
  - 1218.62.32009 Boehringer Ingelheim Investigational Site, Kumtich
  - 1218.62.32005 Boehringer Ingelheim Investigational Site, Massemen-Wetteren
  - 1218.62.32004 Boehringer Ingelheim Investigational Site, Natoye
  - 1218.62.32007 Boehringer Ingelheim Investigational Site, Sint-Job-in't-Goor
  - 1218.62.32002 Boehringer Ingelheim Investigational Site, Tessenderlo
  - 1218.62.32006 Boehringer Ingelheim Investigational Site, Wilsele
- Canada (14):
  - 1218.62.11012 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1218.62.11007 Boehringer Ingelheim Investigational Site, Burnaby, British Columbia
  - 1218.62.11011 Boehringer Ingelheim Investigational Site, St. John's, Newfoundland and Labrador
  - 1218.62.11006 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 1218.62.11001 Boehringer Ingelheim Investigational Site, Barrie, Ontario
  - 1218.62.11003 Boehringer Ingelheim Investigational Site, Brampton, Ontario
  - 1218.62.11004 Boehringer Ingelheim Investigational Site, Markham, Ontario
  - 1218.62.11005 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1218.62.11008 Boehringer Ingelheim Investigational Site, Smiths Falls, Ontario
  - 1218.62.11013 Boehringer Ingelheim Investigational Site, Strathroy, Ontario
  - 1218.62.11014 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1218.62.11010 Boehringer Ingelheim Investigational Site, Charlottetown, Prince Edward Island
  - 1218.62.11002 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1218.62.11009 Boehringer Ingelheim Investigational Site, Point Claire, Quebec
- France (21):
  - 1218.62.3303C Boehringer Ingelheim Investigational Site, Bort-les-Orgues
  - 1218.62.3306A Boehringer Ingelheim Investigational Site, Bourg Des Cptes
  - 1218.62.3303D Boehringer Ingelheim Investigational Site, Bugeat
  - 1218.62.3302H Boehringer Ingelheim Investigational Site, Corsept
  - 1218.62.3308A Boehringer Ingelheim Investigational Site, Derval
  - 1218.62.3302B Boehringer Ingelheim Investigational Site, La Chapelle-sur-Erdre
  - 1218.62.3304A Boehringer Ingelheim Investigational Site, Levallois-Perret
  - 1218.62.3305A Boehringer Ingelheim Investigational Site, Marseille
  - 1218.62.3305B Boehringer Ingelheim Investigational Site, Marseille
  - 1218.62.3305G Boehringer Ingelheim Investigational Site, Marseille
  - 1218.62.3305H Boehringer Ingelheim Investigational Site, Marseille
  - 1218.62.3301A Boehringer Ingelheim Investigational Site, Nantes
  - 1218.62.3302A Boehringer Ingelheim Investigational Site, Nantes
  - 1218.62.3304B Boehringer Ingelheim Investigational Site, Paris
  - 1218.62.3304D Boehringer Ingelheim Investigational Site, Paris
  - 1218.62.3305F Boehringer Ingelheim Investigational Site, Roquevaire
  - 1218.62.3305I Boehringer Ingelheim Investigational Site, Roquevaire
  - 1218.62.3303A Boehringer Ingelheim Investigational Site, Rosiers-d'Égletons
  - 1218.62.3303H Boehringer Ingelheim Investigational Site, Sainte-Fortunade
  - 1218.62.3302I Boehringer Ingelheim Investigational Site, Sautron
  - 1218.62.3302G Boehringer Ingelheim Investigational Site, Vue
- India (5):
  - 1218.62.91001 Boehringer Ingelheim Investigational Site, Bangalore
  - 1218.62.91004 Boehringer Ingelheim Investigational Site, Bangalore
  - 1218.62.91003 Boehringer Ingelheim Investigational Site, Hyderabad, Andra Pradesh
  - 1218.62.91005 Boehringer Ingelheim Investigational Site, Nagpru
  - 1218.62.91002 Boehringer Ingelheim Investigational Site, Trivandrum
- Italy (10):
  - 1218.62.39010 Boehringer Ingelheim Investigational Site, Ancona
  - 1218.62.39006 Boehringer Ingelheim Investigational Site, Catania
  - 1218.62.39004 Boehringer Ingelheim Investigational Site, Genova
  - 1218.62.39009 Boehringer Ingelheim Investigational Site, Gissi (CH)
  - 1218.62.39003 Boehringer Ingelheim Investigational Site, Palermo
  - 1218.62.39001 Boehringer Ingelheim Investigational Site, Pisa
  - 1218.62.39002 Boehringer Ingelheim Investigational Site, Pordenone
  - 1218.62.39012 Boehringer Ingelheim Investigational Site, Ravenna
  - 1218.62.39007 Boehringer Ingelheim Investigational Site, Roma
  - 1218.62.39011 Boehringer Ingelheim Investigational Site, Roma
- Malaysia (5):
  - 1218.62.60002 Boehringer Ingelheim Investigational Site, George Town
  - 1218.62.60001 Boehringer Ingelheim Investigational Site, Kelantan Kota Bahru
  - 1218.62.60005 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 1218.62.60003 Boehringer Ingelheim Investigational Site, Putrajaya
  - 1218.62.60004 Boehringer Ingelheim Investigational Site, Seremban
- Netherlands (8):
  - 1218.62.31007 Boehringer Ingelheim Investigational Site, Almere Stad
  - 1218.62.31004 Boehringer Ingelheim Investigational Site, Breezerveld
  - 1218.62.31005 Boehringer Ingelheim Investigational Site, Etten-Leur
  - 1218.62.31002 Boehringer Ingelheim Investigational Site, Lieshout
  - 1218.62.31001 Boehringer Ingelheim Investigational Site, Oude Pekela
  - 1218.62.31008 Boehringer Ingelheim Investigational Site, Voerendaal
  - 1218.62.31009 Boehringer Ingelheim Investigational Site, Wildervank
  - 1218.62.31003 Boehringer Ingelheim Investigational Site, Woerden
- South Korea (6):
  - 1218.62.82005 Boehringer Ingelheim Investigational Site, Goyang
  - 1218.62.82006 Boehringer Ingelheim Investigational Site, Goyang
  - 1218.62.82003 Boehringer Ingelheim Investigational Site, Incheon
  - 1218.62.82004 Boehringer Ingelheim Investigational Site, Pucheon
  - 1218.62.82002 Boehringer Ingelheim Investigational Site, Seoul
  - 1218.62.82001 Boehringer Ingelheim Investigational Site, Suwon
- Spain (7):
  - 1218.62.34003 Boehringer Ingelheim Investigational Site, Badia Del Vallés (Barcelona)
  - 1218.62.34002 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat (Barcelona)
  - 1218.62.34005 Boehringer Ingelheim Investigational Site, Madrid
  - 1218.62.34006 Boehringer Ingelheim Investigational Site, Madrid
  - 1218.62.34007 Boehringer Ingelheim Investigational Site, Madrid
  - 1218.62.34001 Boehringer Ingelheim Investigational Site, Palma (Mallorca)
  - 1218.62.34008 Boehringer Ingelheim Investigational Site, Palma de Mallorca

REFERENCES:
- [Derived] Ross SA, Rafeiro E, Meinicke T, Toorawa R, Weber-Born S, Woerle HJ. Efficacy and safety of linagliptin 2.5 mg twice daily versus 5 mg once daily in patients with type 2 diabetes inadequately controlled on metformin: a randomised, double-blind, placebo-controlled trial. Curr Med Res Opin. 2012 Sep;28(9):1465-74. doi: 10.1185/03007995.2012.714360. Epub 2012 Aug 13. PMID 22816729

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients treated with matching placebo
- Lina 2.5 Twice Daily (Bid): Patients treated with Linagliptin 2.5mg bid
- Lina 5 Once Daily (qd): Patients treated with Linagliptin 5mg qd
Period: Overall Study
Arm/Group | Placebo | Lina 2.5 Twice Daily (Bid) | Lina 5 Once Daily (qd)
Started | 44 | 223 | 224
Completed | 43 | 207 | 214
Not Completed | 1 | 16 | 10
Not completed — Adverse Event | 0 | 8 | 3
Not completed — Protocol Violation | 0 | 3 | 5
Not completed — Withdrawal by Subject | 0 | 4 | 1
Not completed — Other reason (not specified) | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lina 2.5 Twice Daily (Bid) | Lina 5 Once Daily (qd) | Total
Number analyzed (Participants) | 44 | 223 | 224 | 491
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.9 (10.7) | 58.7 (9.9) | 58.4 (10.6) | 58.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 85 | 103 | 211
  Male | 21 | 138 | 121 | 280
Body Mass Index (BMI) continuous [Mean (Standard Deviation); unit: kg/m^2] | 28.65 (5.53) | 29.77 (5.23) | 29.55 (4.95) | 29.57 (5.13)
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percent] — Baseline HbA1c was determined for the Full Analysis Set with 43 patients treated with Placebo, 214 patients treated with Linagliptin 2.5 bid and 221 patients treated with Linagliptin 5mg qd (478 in total).
  percent | 7.92 (0.74) | 7.96 (0.78) | 7.98 (0.72) | 7.97 (0.75)
Fasting blood plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] — Baseline FPG was determined for the Full Analysis Set (where FPG values were also available) with 41 patients treated with Placebo, 209 patients treated with Linagliptin 2.5 bid and 216 patients treated with Linagliptin 5mg qd (466 in total).
  mg/dL | 166.2 (40.3) | 164.1 (41.8) | 165.8 (35.1) | 165.1 (38.6)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Change From Baseline at Week 12
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 12 HbA1c percent minus the baseline HbA1c percent. Treatment means are adjusted for baseline HbA1c and use of prior oral antidiabetics (OADs) in addition to background metformin.
Time Frame: Baseline and week 12
Population: The Full Analysis Set (FAS) included all treated patients with a baseline and at least one on-treatment HbA1c measurement available. Last observation carried forward (LOCF) was used as the imputation rule.
Measure: Mean (Standard Error); unit: percent
Arm/Group | Placebo | Lina 2.5 Twice Daily (Bid) | Lina 5 Once Daily (qd)
Number analyzed (Participants) | 43 | 214 | 221
percent | 0.28 (0.11) | -0.46 (0.05) | -0.52 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Lina 2.5 Twice Daily (Bid); Linagliptin 2.5mg bid versus Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.74, 95% CI [-0.97 to -0.52], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Placebo vs Lina 5 Once Daily (qd); Linagliptin 5mg qd versus Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.80, 95% CI [-1.02 to -0.58], Standard Error of Mean 0.11
Statistical Analysis 3: Comparison: Lina 2.5 Twice Daily (Bid) vs Lina 5 Once Daily (qd); Linagliptin 2.5mg bid versus Linagliptin 5mg qd; Test type: Non-Inferiority or Equivalence — The pre-defined non-inferiority margin was +0.35; ANCOVA; Mean Difference (Final Values) = 0.06, 95% CI [-0.07 to 0.19], Standard Error of Mean 0.07

2. Secondary Outcome: HbA1c Change From Baseline at Week 6 From Mixed Model Repeated Measures (MMRM) Analysis
Description: Mixed model includes treatment, baseline HbA1c, use of prior oral antidiabetics (OADs) in addition to background metformin, week repeated within patient, week by treatment interaction.
Time Frame: Baseline and week 6
Population: The Full Analysis Set (FAS) included all treated patients with a baseline and at least one on-treatment HbA1c measurement available. No imputation was performed. Patients without a Week 6 value were handled by the statistical model.
Measure: Mean (Standard Error); unit: percent
Arm/Group | Placebo | Lina 2.5 Twice Daily (Bid) | Lina 5 Once Daily (qd)
Number analyzed (Participants) | 43 | 214 | 221
percent | 0.32 (0.08) | -0.34 (0.04) | -0.34 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Lina 2.5 Twice Daily (Bid); Linagliptin 2.5mg bid versus Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.66, 95% CI [-0.83 to -0.48], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: Placebo vs Lina 5 Once Daily (qd); Linagliptin 5mg qd versus Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.66, 95% CI [-0.84 to -0.49], Standard Error of Mean 0.09
Statistical Analysis 3: Comparison: Lina 2.5 Twice Daily (Bid) vs Lina 5 Once Daily (qd); Linagliptin 2.5mg bid versus Linagliptin 5mg qd; Test type: Non-Inferiority or Equivalence — The pre-defined non-inferiority margin was +0.35; Mixed Models Analysis; Mean Difference (Final Values) = 0.00, 95% CI [-0.10 to 0.10], Standard Error of Mean 0.05

3. Secondary Outcome: HbA1c Change From Baseline at Week 12 From Mixed Model Repeated Measures (MMRM) Analysis
Description: as for outcome 2
Time Frame: Baseline and week 12
Population: The Full Analysis Set (FAS) included all treated patients with a baseline and at least one on-treatment HbA1c measurement available. No imputation was performed. Patients without a Week 12 value were handled by the statistical model.
Measure: Mean (Standard Error); unit: percent
Arm/Group | Placebo | Lina 2.5 Twice Daily (Bid) | Lina 5 Once Daily (qd)
Number analyzed (Participants) | 43 | 214 | 221
percent | 0.27 (0.11) | -0.51 (0.05) | -0.55 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Lina 2.5 Twice Daily (Bid); Linagliptin 2.5mg bid versus Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.77, 95% CI [-1.00 to -0.54], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Placebo vs Lina 5 Once Daily (qd); Linagliptin 5mg qd versus Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -0.82, 95% CI [-1.05 to -0.59], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: Lina 2.5 Twice Daily (Bid) vs Lina 5 Once Daily (qd); Linagliptin 2.5mg bid versus Linagliptin 5mg qd; Test type: Non-Inferiority or Equivalence — The pre-defined non-inferiority margin was +0.35; Mixed Models Analysis; Mean Difference (Final Values) = 0.05, 95% CI [-0.08 to 0.18], Standard Error of Mean 0.07

4. Secondary Outcome: FPG Change From Baseline at Week 12
Description: Change from baseline reflects the Week 12 FPG minus the baseline FPG. Treatment means are adjusted for baseline HbA1c, baseline fasting plasma glucose and use of prior oral antidiabetics (OADs) in addition to background metformin.
Time Frame: Baseline and week 12
Population: Patients from FAS with values for FPG at baseline and on-treatment. Last observation carried forward (LOCF) was used as the imputation rule.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Lina 2.5 Twice Daily (Bid) | Lina 5 Once Daily (qd)
Number analyzed (Participants) | 40 | 203 | 213
mg/dL | -3.5 (4.2) | -17.2 (1.9) | -21.3 (1.9)
Statistical Analysis 1: Comparison: Placebo vs Lina 2.5 Twice Daily (Bid); Linagliptin 2.5mg bid versus Placebo; Test type: Superiority or Other; p = 0.0029, ANCOVA; Mean Difference (Final Values) = -13.7, 95% CI [-22.7 to -4.7], Standard Error of Mean 4.6
Statistical Analysis 2: Comparison: Placebo vs Lina 5 Once Daily (qd); Linagliptin 5 mg qd versus Placebo; Test type: Superiority or Other; p = 0.0001, ANCOVA; Mean Difference (Final Values) = -17.8, 95% CI [-26.7 to -8.8], Standard Error of Mean 4.6
Statistical Analysis 3: Comparison: Lina 2.5 Twice Daily (Bid) vs Lina 5 Once Daily (qd); Linagliptin 2.5mg bid versus Linagliptin 5mg qd; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 4.1, 95% CI [-1.0 to 9.2], Standard Error of Mean 2.6 — No non-inferiority margin was pre-defined for FPG

5. Secondary Outcome: FPG Change From Baseline at Week 6 From Mixed Model Repeated Measures (MMRM) Analysis
Description: Mixed model includes treatment, baseline HbA1c, baseline FPG, use of prior oral antidiabetics (OADs) in addition to background metformin, week repeated within patient, week by treatment interaction.
Time Frame: Baseline and week 6
Population: Patients from FAS with values for FPG at baseline and on-treatment. No imputation was performed. Patients without a Week 12 value were handled by the statistical model.
Measure: Mean (Standard Error); unit: percent
Arm/Group | Placebo | Lina 2.5 Twice Daily (Bid) | Lina 5 Once Daily (qd)
Number analyzed (Participants) | 40 | 203 | 213
percent | -1.2 (4.1) | -17.8 (1.9) | -20.1 (1.8)
Statistical Analysis 1: Comparison: Placebo vs Lina 2.5 Twice Daily (Bid); Linagliptin 2.5mg bid versus Placebo; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = -16.6, 95% CI [-25.3 to -7.8], Standard Error of Mean 4.4
Statistical Analysis 2: Comparison: Placebo vs Lina 5 Once Daily (qd); Linagliptin 5mg qd versus Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -18.9, 95% CI [-27.6 to -10.2], Standard Error of Mean 4.4
Statistical Analysis 3: Comparison: Lina 2.5 Twice Daily (Bid) vs Lina 5 Once Daily (qd); Linagliptin 2.5mg bid versus Linagliptin 5mg qd; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 2.3, 95% CI [-2.6 to 7.3], Standard Error of Mean 2.5 — No non-inferiority margin was pre-defined for FPG

6. Secondary Outcome: FPG Change From Baseline at Week 12 From Mixed Model Repeated Measures (MMRM) Analysis
Description: as for outcome 5
Time Frame: Baseline and week 12
Population: as for outcome 5
Measure: Mean (Standard Error); unit: percent
Arm/Group | Placebo | Lina 2.5 Twice Daily (Bid) | Lina 5 Once Daily (qd)
Number analyzed (Participants) | 40 | 203 | 213
percent | -8.7 (5.0) | -18.7 (2.3) | -23.9 (2.2)
Statistical Analysis 1: Comparison: Placebo vs Lina 2.5 Twice Daily (Bid); Linagliptin 2.5mg bid versus Placebo; Test type: Superiority or Other; p = 0.0653, Mixed Models Analysis; Mean Difference (Final Values) = -10.0, 95% CI [-20.6 to 0.6], Standard Error of Mean 5.4
Statistical Analysis 2: Comparison: Placebo vs Lina 5 Once Daily (qd); Linagliptin 5mg qd versus Placebo; Test type: Superiority or Other; p = 0.0047, Mixed Models Analysis; Mean Difference (Final Values) = -15.3, 95% CI [-25.8 to -4.7], Standard Error of Mean 5.4
Statistical Analysis 3: Comparison: Lina 2.5 Twice Daily (Bid) vs Lina 5 Once Daily (qd); Linagliptin 2.5mg bid versus Linagliptin 5mg qd; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 5.3, 95% CI [-0.7 to 11.3], Standard Error of Mean 3.0 — No non-inferiority margin was pre-defined for FPG

7. Secondary Outcome: Percentage of Patients With HbA1c Lowering by 0.5% or More at Week 12
Description: Percentage of patients with HbA1c lowering by at least 0.5% after 12 weeks. The analysis was performed on the full analysis set (FAS) using NCF.
Time Frame: Week 12
Population: The Full Analysis Set (FAS) included all treated patients with a baseline and at least one on-treatment HbA1c measurement available. Patients without a value at Week 12 were analysed as non-responders
Measure: Number; unit: percent
Arm/Group | Placebo | Lina 2.5 Twice Daily (Bid) | Lina 5 Once Daily (qd)
Number analyzed (Participants) | 43 | 214 | 221
percent | 16.3 | 55.1 | 59.7

8. Secondary Outcome: Percentage of Patients With Rescue Therapy
Description: Percentage of patients with rescue therapy at Week 12. The analysis was performed on the full analysis set (FAS) using OC.
Time Frame: 12 weeks
Measure: Number; unit: percent
Arm/Group | Placebo | Lina 2.5 Twice Daily (Bid) | Lina 5 Once Daily (qd)
Number analyzed (Participants) | 43 | 214 | 221
percent | 7.0 | 3.7 | 1.8

9. Secondary Outcome: The Occurrence of a Treat to Target Efficacy Response (HbA1c <7.0%) After 12 Weeks of Treatment
Description: Percentage of those patients with baseline HbA1c >= 7.0% who had HbA1c < 7% at Week 12. The analysis was performed on the full analysis set (FAS) using NCF.
Time Frame: 12 weeks
Population: FAS (NCF) with baseline HbA1c >= 7.0%
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lina 2.5 Twice Daily (Bid) | Lina 5 Once Daily (qd)
Number analyzed (Participants) | 40 | 206 | 215
percentage of participants | 10.0 | 34.0 | 33.0

10. Secondary Outcome: The Occurrence of a Treat to Target Efficacy Response (HbA1c <6.5 %) After 12 Weeks of Treatment
Description: Percentage of those patients with baseline HbA1c >= 6.5% who had HbA1c < 6.5% at Week 12. The analysis was performed on the full analysis set (FAS) using NCF.
Time Frame: 12 weeks
Population: FAS (NCF) with baseline HbA1c >= 6.5%
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lina 2.5 Twice Daily (Bid) | Lina 5 Once Daily (qd)
Number analyzed (Participants) | 43 | 212 | 221
percentage of participants | 0.0 | 12.7 | 11.8

ADVERSE EVENTS:
Time Frame: up to 12 weeks (drug stop) + 7 days (follow-up)
Arm/Group | Placebo | Lina 2.5 Twice Daily (Bid) | Lina 5 Once Daily (qd)
Serious Adverse Events (participants affected / at risk) | 0/44 | 9/223 | 5/224
Other Adverse Events (participants affected / at risk) | 0/44 | 0/223 | 0/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=44) | Lina 2.5 Twice Daily (Bid) (N=223) | Lina 5 Once Daily (qd) (N=224)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Open fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Preoperative care (Surgical and medical procedures) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.